CLINICAL TRIAL: NCT03297619
Title: A Randomized Controlled Trial (RCT) Comparing Acceptance and Commitment Therapy (ACT) and Cognitive Behavioral Therapy (CBT) Self-help Books for Social Anxiety
Brief Title: Self-help Books for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Assistant Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8694
Record Dates: First submitted 2017-09-13; First posted 2017-09-29 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Social Anxiety
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two active self-help interventions for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT self-help book condition (Experimental): Participants in this condition will be assigned to read The Mindfulness and Acceptance Workbook for Social Anxiety and Shyness by Fleming and Kocovski (2013), a self-help book based on acceptance and commitment therapy.
  Interventions: Behavioral: Mindfulness and Acceptance Workbook for Social Anxiety and Shyness
- CBT self-help book condition (Active Comparator): Participants in this condition will be assigned to read The Shyness and Social Anxiety Workbook by Antony and Swinson (2008), a self-help book based on cognitive-behavioral therapy for social anxiety.
  Interventions: Behavioral: The Shyness and Social Anxiety Workbook

INTERVENTIONS:
Behavioral: Mindfulness and Acceptance Workbook for Social Anxiety and Shyness — Participants assigned to this condition will be asked to read this self-help book over an 8-week period.
  Arms: ACT self-help book condition
Behavioral: The Shyness and Social Anxiety Workbook — Participants assigned to this condition will be asked to read this self-help book over an 8-week period (with some chapters omitted).
  Arms: CBT self-help book condition

SUMMARY:
The goal of this study is to compare the efficacy and mechanisms of change of two self-help books for social anxiety in college students in a randomized controlled trial. One book is based on traditional cognitive behavioral therapy and one is based on acceptance and commitment therapy.

This study will test the following hypotheses:

Hypothesis 1: The CBT and ACT book conditions will both experience decreased social anxiety and distress. Life satisfaction and values progress will increase in both conditions.

Hypothesis 2: The CBT condition will result in greater use of reappraisal, the ACT condition will not.

Hypothesis 3: The ACT condition will result in greater use of defusion and decreased psychological inflexibility; the CBT condition will not.

Hypothesis 4: Changes in experiential avoidance and defusion will predict changes in social anxiety and values progress in the ACT condition.

Hypothesis 5: Changes in reappraisal will predict changes in social anxiety in the CBT condition. Change in values progress will be predicted by change in social anxiety in the CBT condition.

Hypothesis 6: The association between social anxiety/negative affect and values progress will decrease or disappear in the ACT condition (i.e., decoupling), and remain the same in the CBT condition.

DETAILED DESCRIPTION:
The investigators aim to recruit 100 participants for this RCT (50 per treatment condition). This will provide adequate power (0.80) to detect differences between groups of medium effect size (d=0.50). Eligibility criteria will include being 18 years of age or older, being a current Utah State University (USU) student, not having participated in previous self-help studies conducted by the USU Contextual Behavioral Science (CBS) Lab, being interested in self-help for social anxiety, and scoring at least a 6 on the Mini-SPIN, a screener for social anxiety symptoms. Participants will be recruited via SONA, flyers, online postings, classroom announcements, and through a general online screener for various USU CBS Lab studies.

Total study participation will occur over approximately 8 weeks. All study procedures will be completed online, on a computer/mobile phone. After completing informed consent, participants will complete a baseline survey.

At the end of the baseline survey, participants will be randomly assigned to use a book based on CBT (The Shyness and Social Anxiety Workbook) or on ACT (The Mindfulness and Acceptance Workbook for Social Anxiety and Shyness). Note that participants will be asked not to access other self-help books during the study duration. Participants will be provided with an 8-week reading schedule and a link to the assigned book. Participants will be asked to complete a midtreatment survey 4 weeks after the beginning of treatment. The midtreatment survey will include questions about adherence. Participants will be asked to complete a posttreatment survey 8 weeks after the beginning of treatment. This survey will also ask about adherence (reading, use of strategies taught in the book, and exposures). Researcher contact will involve reminders to complete assessments, a basic email assistance in identifying and responding to any barriers to using the self-help book, and twice-weekly reminders of the suggested reading schedule.

After completing the initial assessment participants will be sent a link to The Mindfulness and Acceptance Workbook for Social Anxiety and Shyness if they are assigned to the ACT condition, or a link to the Shyness and Social Anxiety Workbook if they are in the CBT condition. They will be able to access the book online at any time. Participants will be asked to read assigned chapters on an 8-week schedule.

The primary treatment components in the Mindfulness and Acceptance Workbook for Social Anxiety and Shyness are psychoeducation, values and goals, mindfulness, acceptance, defusion, and committed action. The book uses writing exercises to identify patterns/values/goals/committed action, guided and unguided mindfulness meditations, and acceptance exercises.

The primary treatment components in The Shyness and Social Anxiety Workbook are psychoeducation (introducing the cognitive behavioral model), self-assessment (e.g., anxiety hierarchy, identifying beliefs, identifying avoidance), cognitive restructuring, situational exposure, exposure to physical symptoms, and maintenance/consolidation. The book also includes a chapter on motivation and treatment options and a chapter on medication, but these were omitted in a previous trial of the book and will also be omitted in the present study. There is also a chapter on social skills, which will be omitted in order to keep dosage similar between the two books. The book briefly mentions acceptance in the context of exposure (e.g., fear will stick around longer after fighting it) but includes no major acceptance or mindfulness components.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Enrolled at Utah State University
* Have not participated in other self-help studies run by the USU CBS Lab
* Interested in using self-help book for social anxiety
* Scoring at least a 6 on the Mini Social Phobia Inventory (Mini-SPIN), a validated social anxiety screening measure

Exclusion Criteria:

* Exclusion criteria mirror inclusion criteria: below the age of 18, not a student at Utah State University, have participated in previous self-help studies run by the CBS Lab, not interested in using a self-help book for social anxiety, or scoring a 5 or lower on the Mini-SPIN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale - Self Report (Fresco et al., 2001) | Posttreatment (9 weeks after baseline)
  A self-report measure of fear and avoidance of social situations.

SECONDARY OUTCOMES:
General Health Questionnaire-12 (Banks et al., 1980; Goldberg, 1978) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of overall psychological distress.
Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Social Roles And Activities Short Form 8 v2.0 (Hahn et al., 2014) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of social functioning
Valuing Questionnaire - Progress subscale (Smout, Davies, Burns, & Christie, 2014) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of progress toward personal values.

OTHER OUTCOMES:
Believability of Anxious Feelings and Thoughts Questionnaire (Herzberg et al., 2012) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of cognitive fusion as it relates to anxiety.
Cognitive Fusion Questionnaire (Gillanders et al., 2014) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of overall cognitive fusion.
Appraisal of Social Concerns Scale (Telch et al., 2004) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  A self-report measure of concern regarding negative social outcomes.
Reappraisal and mindfulness items (Goldin, Morrison, Jazaieri, Heimberg, & Gross, 2017) | Baseline, midtreatment (5 weeks after baseline), and posttreatment (9 weeks after baseline)
  These items will be used to measure use of cognitive reappraisal and mindful acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Connor KM, Kobak KA, Churchill LE, Katzelnick D, Davidson JR. Mini-SPIN: A brief screening assessment for generalized social anxiety disorder. Depress Anxiety. 2001;14(2):137-40. doi: 10.1002/da.1055. PMID 11668666
- [Background] Antony, M. M., & Swinson, R. P. (2008). The shyness and social anxiety workbook. Oakland, CA: New Harbinger Publications, Inc.
- [Background] Fleming, J. E., & Kocovski, N. L. (2013). The mindfulness and acceptance workbook for social anxiety and shyness. Oakland, CA: New Harbinger Publications, Inc.
- [Background] Abramowitz JS, Moore EL, Braddock AE, Harrington DL. Self-help cognitive-behavioral therapy with minimal therapist contact for social phobia: a controlled trial. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):98-105. doi: 10.1016/j.jbtep.2008.04.004. Epub 2008 Apr 26. PMID 18514614
- [Background] Fresco DM, Coles ME, Heimberg RG, Liebowitz MR, Hami S, Stein MB, Goetz D. The Liebowitz Social Anxiety Scale: a comparison of the psychometric properties of self-report and clinician-administered formats. Psychol Med. 2001 Aug;31(6):1025-35. doi: 10.1017/s0033291701004056. PMID 11513370
- [Background] Banks, M. H., Clegg, C. W., Jackson, P. R., Kemp, N. J., Stafford, E. M., & Wall, T. D. (1980). The use of the General Health Questionnaire as an indicator of mental health in occupational studies. Journal of Occupational Psychology, 53, 187-194.
- [Background] Goldberg, D. (1978). Manual of the GHQ. Windsor: NFER.
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the Valuing Questionnaire (VQ). Journal of Contextual Behavioral Science, 3, 164-172. http://doi.org/10.1016/j.jcbs.2014.06.001
- [Background] Herzberg KN, Sheppard SC, Forsyth JP, Crede M, Earleywine M, Eifert GH. The Believability of Anxious Feelings and Thoughts Questionnaire (BAFT): a psychometric evaluation of cognitive fusion in a nonclinical and highly anxious community sample. Psychol Assess. 2012 Dec;24(4):877-91. doi: 10.1037/a0027782. Epub 2012 Apr 9. PMID 22486595
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Schultz LT, Heimberg RG, Rodebaugh TL, Schneier FR, Liebowitz MR, Telch MJ. The appraisal of social concerns scale: psychometric validation with a clinical sample of patients with social anxiety disorder. Behav Ther. 2006 Dec;37(4):392-405. doi: 10.1016/j.beth.2006.06.001. Epub 2006 Aug 4. PMID 17071216
- [Background] Telch MJ, Lucas RA, Smits JA, Powers MB, Heimberg R, Hart T. Appraisal of social concerns: a cognitive assessment instrument for social phobia. Depress Anxiety. 2004;19(4):217-24. doi: 10.1002/da.20004. PMID 15274170
- [Background] Goldin PR, Morrison AS, Jazaieri H, Heimberg RG, Gross JJ. Trajectories of social anxiety, cognitive reappraisal, and mindfulness during an RCT of CBGT versus MBSR for social anxiety disorder. Behav Res Ther. 2017 Oct;97:1-13. doi: 10.1016/j.brat.2017.06.001. Epub 2017 Jun 3. PMID 28654771